CLINICAL TRIAL: NCT07003932
Title: Remote Monitoring After Total Knee Replacement
Acronym: OA-AID TKR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Anne Therese Tveter, Professor, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 855137
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Knee Arthroplasty, Total
Keywords: knee arthroplasty; remote follow-up; non-inferiority
MeSH Terms: interventions — Remote Patient Monitoring

STUDY DESIGN:
Intervention Model Description: Randomized, open-labeled, parallel group, non-inferiority, single-site clinical trial
Masking Description: The statistician conducting the primary analysis will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients randomly allocated to standard follow-up will be summoned for a hospital visit with a physiotherapist at 8 weeks and 12 months post-surgery. The physiotherapist will conduct an assessment in line with regular clinical practice. If the patient is experiencing lack of improvement or adverse events, an orthopedic surgeon may be consulted. The patients will also answer patient-reported outcomes at 8 weeks and 6- and 12 months post-surgery, however, these answers will not be monitored.
  Interventions: Other: Usual Care
- Remote monitoring (Experimental): Patients randomly allocated to the remote monitoring group will answer patient-reported outcome at 1, 2, 3, 6 and 12 months. They will be provided with a brief introduction from the study personnel on how to answer questions remotely through the Youwell platform. Patients will get an SMS notification on their mobile phone with a link to the questionnaire. They will have to log in with BankID to access the questionnaire. A physiotherapist will monitor the answers and will contact the patient if an unexpected deterioration or adverse events are detected.
  Interventions: Other: Remote monitoring

INTERVENTIONS:
Other: Remote monitoring — The remote monitoring group will be more closely followed than the control group in order to detect any deterioration over time. This group will not be scheduled for a face-to-face consultation unless it is deemed necessary by a physiotherapist or if the patient contacts the hospital themselves.
  Arms: Remote monitoring
Other: Usual Care — The control group will follow usual care with face-to-face consultation with a physiotherapist at 2 and 12 months. They will also anwer questionnaires at 2, 6 and 12 months, but these will not be monitored.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to evaluate the effect, cost-effectiveness, safety and satisfaction with replacing standardized, pre-scheduled face-to-face visits with remote monitoring and video consultations or face-to-face consultations only when needed after total knee replacement surgery due to knee osteoarthritis.

The primary outcome is the probability of being a OMERACT-OARSI responder at 6 months post-surgery. This is a composite index where participants are classified as a responder or non-responder based on improvement in pain, function and/or disease activity. Health-related quality of life and healthcare costs will be used to determine cost-effectiveness. Patient-reported adverse events and statisfaction will be used to determine safety and satisfaction.

Patients will be recruited from Diakonhjemmet Hospital. Patients undergoing total knee replacement surgery will be randomly allocated to a control group who are summoned for a face-to-face consultation at Diakonhjemmet Hospital at 2 and 12 months, or a remote monitoring group who will not be scheduled for hospital visits but will answer patient-reported outcomes throught a web-application at 1, 2, 3, 6 and 12 months post-surgery and only be scheduled for hospital visits when needed.

An additional study with follow-up after 5 and 10 years will be conducted.

DETAILED DESCRIPTION:
Participants are eligible for inclusion in the study if the following criteria apply:

* men and women, 50 years of age or older
* referred to total knee replacement surgery due to knee osteoarthritis

Participants are excluded from the study of any of the following criteria apply:

* revision of previous total knee replacement surgery
* serious comorbidities (such as severe malignancues, severe diabetes mellitus, severe infections, uncontrollable hypertension, severe cardiovascular disease, severe respiratory disease)
* congnitive dysfunction
* total knee replacement surgery due to trauma or inflammatory joint disease (such as psoriatic arthritis or rheumatoid arthritis)
* unable to understand Norwegian
* Cannot answer questionnaires digitally (lack BankID, do not possess a smartphone
* deemed inappropriate for remote monitoring by orthopedic surgeon

Patients included in both treatment arms will receive medical treatment according to current treatment recommendations as applied by the treating orthopedic surgeon after total knee replacement. All partients are recommended to seek physiotherapy treatment in primary care after surgery

Patients randomly allocated to the control group will be summoned for a hospital visit with a physiotherapist at 2 and 12 months. The physiotherapist will conduct assessment in line with regular clinical practice. If the patient is experiencing lack of improvement or adverse events, an orthopedic surgeon may be consulted. The patients will also answer patient-reported outcomes at 8 weeks and 6- and 12 months post-surgery, however, these answers will not be monitored.

Patients randomly allocated to the remote monitoring group will answer patient-reported outcome at 1, 2, 3, 6 and 12 months. They will be provided with a brief introduction from the study personnel on how to answer questions remotely through the Youwell platform. Patients will get an SMS notification on their mobile phone with a link to the questionnaire. They will have to log in with BankID to access the questionnaire. A physiotherapist will monitor the answers and will contact the patient if an unexpected deterioration or adverse events are detected.

Data will be collected through Nettskjema or the Youwell software program and will be stored in Services for Sensitive Data (TSD) and a a secure server at Diakonhjemmet Hospital.

The following data will be recorded through self-report in the baseline questionnaire:

* Demography: mobile number, education, work status, living arrangement, socioeconomic status, social support, expectations about treatment, fear of movement, catastrophizing, self-efficacy
* Disease variables: KOOS, other joints with osteoarthritis, duration of complaint, previous treatment, fatigue, disease activity, pain, function, pain medication, osteoarthritis quality indicators, knee flexion/extension, use of walking aids
* Lifestyle variables: physical activity, motivation for exercise, motivation for surgery
* Health competency, digital self-efficacy
* Patient satisfaction
* Health-related quality of life The following information will be collected from medical records
* Demographic variables: Age, gender, height, weight, comorbidity, referred knee, smoking,
* General medical history: description of radiographs, type of scheduled arthroplasty, joint status prior to surgery

Patients allocated to the remote monitoring group will receive an SMS with link to questionnaires in the Youwell platform at 1, 2, 3, 6 and 12 months. The following data will be collected for the remote monitoring group:

* Global rating of change
* Pain/Pain medication
* Fear of movement
* Expectations about treatment
* Disease activity
* Signs inflammation/swelling
* Function/activity
* Knee flexion/extension
* Use of walking aids
* Exercise
* Contact with physiotherapist/ rehabilitation stay
* Adverse events
* Patient satisfaction with care

A highly experienced physiotherapist will review the answers and based on these make a clinical judgement whether there is a need to call the patient or summon the patient for a physical examination, or if the patient seems to manage well at home.

Patients in the control group will also answer the remote monitoring questionnaire at 2 months, however, their answers will not be monitored (just for research purposes).

At follow-up, the following variables will be collected:

* Global rating of change
* Disease variables: KOOS, fatigue, disease activity, pain, function, pain medication,
* Fear of movement
* Self-efficacy
* Knee flexion/extension
* Lifestyle variables: physical activity,
* Patient satisfaction with care
* Health-related quality of life
* Health care costs: hospital stay, rehabilitation stay, travel distance to hospital, transportation, health care use
* Adverse events

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 50 years of age or older
* Reffered to total knee replacement surgery due to knee osteoarthritis

Exclusion Criteria:

* Revision of previous total knee replacement surgery
* Serious comorbidities (such as severe malignancies, severe diabetes mellitus, severe infections, uncontrollable hypertension, severe cardiovascular disease, severe respiratory disease)
* Congitive dysfunction
* Total knee replacement surgery due to trauma or inflammatory joint disease (such as psoriatic arthritis or rheumatoid arthritis)
* Unable to understand Norwegian
* Low digital competency/ cannot answer questionnaires digitally (lack BankID, do not possess a smartphone)
* Deemed inappropriate for remote monitoring by orthopedic surgeon

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
OMERACT-OARSI responder criteria | Baseline, 6 months
  The OMERACT-OARSI responder criteria is a composite index where participants are classifies as responders or non-responders (binary outcome) based on the following criteria:
  High improvement on pain or function
  * ≥50% improvement + absolute change of ≥2 points in pain, OR
  * ≥50% improvement + absolute change of ≥2 point on KOOS) OR Improvement in at least two of the three following
  * ≥20% improvement + absolute change of ≥1 point in pain
  * ≥20% improvement + absolute change of ≥1 point in function
  * ≥20% improvement + absolute change of ≥1 point in disease activity

SECONDARY OUTCOMES:
OMERACT-OARSI responder criteria | Baseline, 12 months
  The OMERACT-OARSI responder criteria is a composite index where participants are classifies as responders or non-responders (binary outcome) based on the following criteria: High improvement on pain or function • ≥50% improvement + absolute change of ≥2 points in pain, OR • ≥50% improvement + absolute change of ≥2 point on KOOS) OR Improvement in at least two of the three following • ≥20% improvement + absolute change of ≥1 point in pain • ≥20% improvement + absolute change of ≥1 point in function • ≥20% improvement + absolute change of ≥1 point in disease activity
Healthcare costs | Baseline, 6 and 12 months
  Direct (consultations in primary or specialist healthcare) and indirect costs (sick leave, medication, travel costs) collected from national registers (NAV, KUHR, NPR) or self-report. Summed up to cost per patient (euro).
Health-related quality of life (EQ5D-5L) | Baseline, 6 months, 12 months
  5 dimensions rated on a 5-point Likert scale, calculated utility score between 0 and 1 (best health)
Safety measures | 1 month, 2 months, 3 months, 6 months, 12 months
  Any adverse events during the follow-up period. Any contact with hospital, emergency unit and general practitioned due to acute worsening. 1 and 3 months only for the remote monitoring group
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 6 months, 12 months
  Assessment of three dimentions of the KOOS (pain, activity in daily living and health-related quality of life) summed up to 0-100 scales where 100 is best score.
Change in pain | Baseline, 2 months, 6 months, 12 months
  Measured on numeric rating scales (0-10) with higher score indicating more pain
Change in disease activity | Baseline, 2 months, 6 months, 12 months
  Measured on a numeric rating scale (0-10) with 10 indicating worst disease activity.
Satisfaction with care | 2 months, 6 months, 12 months
  Measured on a numeric rating scale (0-10) with higher score indicating higher satisfaction with care.
Satisfaction with total knee replacement surgery | 2 months, 6 months, 12 months
  Assessed using 4 primary questions, each rated on a 5-point Likert scale (from "very satisfied" to "very dissatisfied"), and a question about change in health-related quality of life rated on a 6-point scale (from "more improvement than I ever dreamed about" to "the quality of my life is worse")
Change in range of motion | Baseline, 1, 2, 3, 6, 12 months
  Knee flexion and extension is self-reported based on pictures of different degrees of range of motion. Measurement at 1 and 3 months only for the remote monitoring group.
Number of extra visits | Baseline to 12 months
  Number of extra visits in both groups

OTHER OUTCOMES:
Fatigue | Baseline, 2 months, 6 months, 12 months
  Measured on a numeric rating scale (0-10) with 10 indicating most fatigue
Change in problems related to daily activity | Baseline, 2 months, 6 months, 12 months
  Measured on a numeric rating scale (0-10) with 10 indicating more problems (question no.6 in the WPAI questionnaire)
Pain self-efficacy Questionnaire (PSEQ-2) | Baseline, 2 months, 6 months, 12 months
  Two questions on pain self-efficacy measured on a 6-point scale (not at all confident to completely confident)
OsteoArthritis Quality Indicator questionnaire | Baseline
  17 item quality indicator questionnaire with yes, no, don't know/not relevant response categories. Summarized to a pass rate (number of yes divided by number of yes+number of no responses)
Motivation for knee exercises | Baseline
  Measured on a numeric rating scale from 0 to 10, with 10 indicating highly motivated for exercising.
Motivation for knee surgery | Baseline
  Measured on a numeric rating scale from 0 to 10, with 10 indicating highly motivated for undergoing knee surgery
Self-reported exercise | Baseline, 2 months, 6 months, 12 months
  Measured with a question on how often the individual exercise with increased breathing and heart rate for at least 30 minutes. With five response categories (3 times or more per week; 1-2 times per week; 1-2 times per month; do not exercise regularily; cannot exercise)
Global rating of change in the knee | 2 months, 6 months, 12 months
  One question with five response categories asking about experience of change in the knee. Responses from "a very small degree" to "a very large degree"
Digital self-efficacy | Baseline
  Six questions measuring how well the patients manage smartphones, padlets, pc, apps, and login with BankID and Helsenorge.no. Answered on a 5-point scale fron very poorly to very good, with an additional option of "never tried"
Demographics | Baseline
  Questions about age, gender, hight, weight, education level, working status, living arrangements, smoking, comorbidities.
Joint-spesific measures | Baseline
  Questions related to referred joint, other joints with pain/problems
Current treatment | Baseline, 1, 2, 3, 6 and 12 months
  Questions about if and how often they have been visiting a physiotherapist
  (1 and 3 months only for the remote monitoring group)
Satisfaction with follow-up | 6 and 12 months
  Measured on a five-point Likert scale, from "very satisfied" to "very dissatisfied"
Usability of remote follow-up | 6 and 12 months
  Measured with two questions from the system usability scale, modified to this study. The questions focus on the ease of answering the questionnaires and if help was needed. Measured on a 5-point likert scale from "totally disagree" to "totally agree"
Adherence to answering remote monitoring questionnaire | 1, 2, 3, 6 and 12 months
  Number of remote monitoring questionnaires answered (1, 2, 3, 6 and 12 months)
Previous treatment | Baseline
  Reporting of previous treatment (physiotherapy, osteoarthritis seminars, previous surgery in referred knee, previous arthroplasty in opposite knee)
Socioeconomic status | Baseline
  Reporting of sosioeconomic status and if they have someone to help if needed
Change in use of medication | 1, 2, 3 and 6 months
  Self-reported change in medication use (1 and 3 months only for remote monitoring group)
Fear of movement | Baseline, 1, 2, 3 months
  Measured on a 7-point likert scale, measurement at 1 and 3 months only for the remote monitoring group. Response categories from "totally disagree" to "totally agree"
Health competency | Baseline
  Measured on a 5-point likert scale, related to the understanding of their osteoarthritis disease and the treatment of their disease. Response categories from "completely" to "not at all"
Expectations about treatment | Baseline
  Measured with two questions from the Standford Expectations of Treatment Scale, focusing on expectations about the result of surgery. In addition, one question about expectancy of improvement with exercise. All measured on 7-point likert scales, from "totally disagree" to "totally agree".

CONTACTS AND LOCATIONS:
Locations (1):
- Diakonhjemmet Hospital, Oslo, Please Select, Norway

IPD SHARING:
Plan to Share IPD: No
Due to GDPR regulations, IPD cannot be shared